CLINICAL TRIAL: NCT07258121
Title: A Phase 1/2 Dose Escalation and Cohort Expansion Study of the Tolerability, Safety, Efficacy, and Pharmacokinetics of ZGGS34 in Participants With Advanced Solid Tumors
Brief Title: Study of ZGGS34 in Participants With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZGGS34-001
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): A rapid titration followed by the traditional "3 + 3" design will be used for dose escalation: rapid titration is applied to the first cohort, and the conventional "3 + 3" method is used for all subsequent cohorts. Dose escalation is planned to proceed through the following dose levels: 0.5 mg, 1.5 mg, 5.0 mg, 15.0 mg, 30.0 mg, 60.0 mg, and 100.0 mg. The initial dosing frequency is set at once every two weeks (Q2W).
  Interventions: Biological: ZG006
- Part 2: Dose Expansion (Experimental): Based on the RP2D identified in the Part 1 dose-escalation study of ZGGS34, expansion cohorts will be enrolled distinct solid-tumor populations to further evaluate the preliminary efficacy and safety of the selected ZGGS34 monotherapy dose.
  Interventions: Biological: ZG006

INTERVENTIONS:
Biological: ZG006 — ZG006 will be administered as an intravenous (IV) infusion.

SUMMARY:
This is a multicenter, open-label Phase 1/2 study in participants with advanced solid tumors. The study consists of two parts: Part 1 is a dose-escalation phase to evaluate the safety and tolerability of ZGGS34 in advanced solid tumor participants; Part 2 is a cohort-expansion phase to assess the efficacy and safety of ZGGS34 (± chemotherapy) in selected MUC17-positive advanced solid tumor participants.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form;
* Male or female 18~75 years old.
* Archived tumor tissue within 24 months or fresh biopsy specimens must be provided for detection of MUC17 expression, and with positive MUC17 results required.
* Subjects in different study parts need to meet the following requirements:

Part 1: Dose Escalation Study： Histologically or cytologically confirmed advanced solid tumors who have failed standard treatment or no standard treatment available, or were intolerant to standard treatments.

Part 2: Cohort Expansion Study： Cohort 1 (Gastric cancer): Previously received at least one line systematic treatment and failed; HER2 status negative; Cohort 2 (Pancreatic cancer): Previously received at least one line systematic treatment and failed; Cohort 3 (Colorectal cancer): Previously received at least one line systematic treatment and failed; If patients with MSI-H/dMMR, prior PD-1 therapy is required. Cohort 4: Other patients with advanced solid tumors who have failed standard treatment or have no standard treatment available.

Exclusion Criteria:

* Patients having received any of the following treatments:

Prior combination or sequential use of drugs targeting anti-MUC17 (including investigational drugs);Chemotherapy, immunotherapy, targeted therapy, endocrine therapy, and biological targeted medicines ≤ 4 weeks before the first dose. Local palliative radiotherapy and a small molecule targeted therapy ≤ 2 weeks before the first dose; Systemic immunosuppressive medications, such as corticosteroid within 14 days prior to the first dose; Use of any live or live attenuated vaccines against viral infections within 4 weeks of first dose.

* The investigator considers the subject unsuitable for enrollment in this clinical study for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity (DLT) | Up to 28 days
Incidence of Treatment-emergent adverse events (TEAEs) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Principal Investigator — Henan Cancer Hospital